CLINICAL TRIAL: NCT01995383
Title: A Single Oral Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO6836191 in Healthy Male Subjects Including a Single Intravenous Microdose of RO6836191
Brief Title: A Single Ascending Dose Study Investigating the Safety, Pharmacokinetics and Pharmacodynamics of RO6836191 in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: WP28586
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Part 1: Placebo (PL) (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 1: Single Ascending Doses (SAD) of RO6836191 (Experimental)
  Interventions: Drug: RO6836191
- Part 2: PL: Low-salt (LS) followed by normal-salt (NS) diet (Placebo Comparator)
  Interventions: Other: LS followed by NS diet condition; Drug: Placebo; Drug: RO6836191
- Part 2: PL: NS followed by LS diet (Placebo Comparator)
  Interventions: Other: NS followed by LS diet condition; Drug: Placebo; Drug: RO6836191
- Part 2: RO6836191: LS followed by NS diet (Experimental)
  Interventions: Other: LS followed by NS diet condition; Drug: RO6836191
- Part 2: RO6836191: NS followed by LS diet (Experimental)
  Interventions: Other: NS followed by LS diet condition; Drug: RO6836191

INTERVENTIONS:
Other: LS followed by NS diet condition — LS diet period followed by NS diet period
  Arms: Part 2: PL: Low-salt (LS) followed by normal-salt (NS) diet; Part 2: RO6836191: LS followed by NS diet
Other: NS followed by LS diet condition — NS diet period followed by LS diet period
  Arms: Part 2: PL: NS followed by LS diet; Part 2: RO6836191: NS followed by LS diet
Drug: Placebo — Single oral administrations
  Arms: Part 1: Placebo (PL)
Drug: Placebo — 2 single oral administrations
  Arms: Part 2: PL: Low-salt (LS) followed by normal-salt (NS) diet; Part 2: PL: NS followed by LS diet
Drug: RO6836191 — Orally administered, single ascending doses
  Arms: Part 1: Single Ascending Doses (SAD) of RO6836191
Drug: RO6836191 — 2 single oral doses
  Arms: Part 2: RO6836191: LS followed by NS diet; Part 2: RO6836191: NS followed by LS diet
Drug: RO6836191 — Intravenous administration
  Arms: Part 2: PL: Low-salt (LS) followed by normal-salt (NS) diet; Part 2: PL: NS followed by LS diet; Part 2: RO6836191: LS followed by NS diet; Part 2: RO6836191: NS followed by LS diet

SUMMARY:
This single-center, randomized, placebo-controlled, double-blind study will assess the safety, pharmacokinetics and pharmacodynamics of RO6836191 in healthy male volunteers in two parts. Part 1 will assess the safety of oral single ascending doses of RO6836191 compared to placebo in fasted volunteers. In Part 2, participants will be given two single oral doses of RO6836191 or placebo under low or normal-salt diet conditions. A subset of these participants will subsequently receive a single IV dose of RO6836191 for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, aged 18 to 45 years old.
* No active or chronic disease following a detailed medical and surgical history and complete physical examination.
* A BMI between 18 to 30 kg/m2 inclusive.
* Use of a highly effective form of birth control for the duration of the study and until 90 days after the last dose.

Exclusion Criteria:

* Any clinically relevant current or history of conditions or illnesses.
* Clinically significant symptoms of infection within 5 days of the first dosing day or a history of recurrent infections.
* Any suspicion or history of alcohol abuse and/or consumption of other drugs of abuse.
* Smokers unable or unwilling to restrict to 5 cigarettes daily during the study and to not smoke during the stay at the clinic.
* Any cardiac abnormalities.
* Blood donation over 450 mL within three months prior to screening.
* Participation in an investigational drug or device study within 3 months prior to dosing.
* Corticosteroid use within 3 months prior to dosing.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Part 2: Area under the concentration-time curve (AUC) | Up to Day 35
Part 2: Plasma aldosterone levels | Up to 2 days after drug administration
Part 2: Urine aldosterone levels | Up to 3 days after drug administration
Part 1: Plasma aldosterone levels | Up to Day 5
Part 1: Urine aldosterone levels | Up to Day 3
Part 2: Incidence of AEs | Up to 12 weeks
Parts 1: Incidence of adverse events (AE) | Until Day 21

SECONDARY OUTCOMES:
Part 2: Volume of distribution after intravenous administration | Days 28-37

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Marlton, New Jersey, United States

REFERENCES:
- [Derived] Bogman K, Schwab D, Delporte ML, Palermo G, Amrein K, Mohr S, De Vera Mudry MC, Brown MJ, Ferber P. Preclinical and Early Clinical Profile of a Highly Selective and Potent Oral Inhibitor of Aldosterone Synthase (CYP11B2). Hypertension. 2017 Jan;69(1):189-196. doi: 10.1161/HYPERTENSIONAHA.116.07716. Epub 2016 Nov 21. PMID 27872236